CLINICAL TRIAL: NCT05272137
Title: Prospective Data Collection to Evaluate the Feedback Control of the Saluda Medical's Evoke Spinal Cord Stimulation System in the Treatment of Patients With Chronic Pain of the Trunk and/or Limbs
Brief Title: Evoke Data Collection Study Germany
Status: Completed | Type: Observational
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: D100967
Record Dates: First submitted 2022-01-13; First posted 2022-03-09 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECAP-controlled, closed-loop SCS: Spinal cord stimulation that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude
  Interventions: Device: Evoke Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Evoke Spinal Cord Stimulation (SCS) System — A spinal cord stimulation system that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude

SUMMARY:
The objective of this multicentre study is to collect electrophysiological and device data from the Evoke Closed-Loop SCS system in the treatment of chronic pain of the trunk and/or limbs, in a real world setting under normal conditions of use.

ELIGIBILITY:
Inclusion Criteria:

* Patient approval for data collection and transfer of de-identified data to sponsor.

Exclusion Criteria:

* No further exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients, age ≥ 18 years, suffering from chronic pain in the trunk and/or limbs, whom are implanted with the Saluda Medical Evoke SCS system.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
ECAP Measurement in Microvolts | through 6 months post-implant
  Evoked Compound Action Potentials (ECAPs) as a measure of spinal cord activation

CONTACTS AND LOCATIONS:
Locations (1):
- Universität Düsseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nijhuis H, Kallewaard JW, van de Minkelis J, Hofste WJ, Elzinga L, Armstrong P, Gultuna I, Almac E, Baranidharan G, Nikolic S, Gulve A, Vesper J, Dietz BE, Mugan D, Huygen FJPM. Durability of Evoked Compound Action Potential (ECAP)-Controlled, Closed-Loop Spinal Cord Stimulation (SCS) in a Real-World European Chronic Pain Population. Pain Ther. 2024 Oct;13(5):1119-1136. doi: 10.1007/s40122-024-00628-z. Epub 2024 Jul 2. PMID 38954217